CLINICAL TRIAL: NCT02366104
Title: Brasília Study on Healthy Aging
Acronym: BSHA
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Instituto de Cardiologia Biocardios (Unknown); University of Brasilia (Other)
Responsible Party: Principal Investigator, Andrei Carvalho Sposito, M.D., Ph.D., University of Campinas, Brazil
Other Study IDs: Gerus
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: Cardiovascular Diseases; Aged; Primary Prevention
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma Leukocyte DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
BSHA is a cohort study of healthy elderlies enrolled voluntarily. It has been ongoing since December 2008. And the purpose of this study is to assess clinical and biological markers of cardiovascular risk in very elderly participants.

DETAILED DESCRIPTION:
Non-institutionalized outpatients under preventive care were voluntarily enrolled into the study. Participants were aged of 80 years or over, have never manifested myocardial infarction, stroke or peripheral arterial disease. Enrolled participants underwent a detailed clinical examination, including assessment of anthropometric measures, quality of life by the WHOQOL-BREF, psychological test by Geriatric Depression Scale (GDS) and cognitive function by the mini-mental state examination (MMSE). After 12h of overnight fasting, the study participants underwent to blood sampling collection for biochemical analysis and freezing of plasma, serum and DNA. Immediately after blood collection, participants underwent to cardiovascular ultrasound evaluations and computed tomography (CT) scans during the week following the initial assessment. After baseline measurements, all participants were referred to the study as outpatient clinic for prospective medical follow-up evaluations.

Anthropometric measures: body weight, height, waist circumference and skinfold thickness (triceps, biceps, suprailiac and subscapular) were measured. Body mass index (BMI) was calculated. Skinfold thickness was the mean of triplicate measurements at the right side, using a skinfold caliper (WCS Plus®, Cardiomed, Curitiba, Brazil).

Biochemical analysis: After collection, EDTA blood was centrifuged at 5 ◦ C, 4500 rpm for 15min to separate plasma and carrying out the following measurements: glucose (Glucose GOD-PAP, Roche Diagnostics, Mannheim, USA), total cholesterol (CHOD-PAP, Roche Diagnostics, Mannheim, USA), triglycerides (GPO-PAP, Roche Diagnostics, Mannheim, USA), HDL-C (HDL cholesterol without pretreatment, Roche Diagnostics, Mannheim, USA), C-reactive protein (highly sensitive, CardioPhase, Dade Behring, Marburg, USA), urea and creatinine (GLDH, Hitachi, Tokyo, Japan), fibrinogen (Sysmex CA 1500, Siemens, Munich, Germany), interleukin (IL) 10 and tumor necrosis factor type alpha (TNF-alpha) (eBioscience, San Diego, CA, USA). Parathyroid hormone (PTH) and calcitonin (Immulite 2000, Siemens, Los Angeles, CA, USA), bone fraction of alkaline phosphatase (Hitachi Autoanalyzer, Tokyo Japan), calcium (Hitachi Autoanalyzer, Tokyo, Japan), apoA and apoB (Behring Nephelometer BNII, Dade Behring, Marburg, Germany) were also measured.

Carotid ultrasound: The evaluation of intima-media thickness (IMT) and presence of carotid plaques were assessed using high-resolution B-mode ultrasound (Philips, model IE 33, 3-9 MHz linear transducer, Philips Medical Systems, Andover, MA, USA) according to the protocols of the American Association of Echocardiography. Bilateral measurements were made at the posterior wall of the bulb of the common carotid artery and at the internal carotid artery through a program of automatic edge detection (QLAB version 6.0 software). Carotid plaque was defined as the presence of focal thickening of at least 50% higher than surrounding areas or as focal region with IMT > 1.5 mm and distinct adjacent edges.

Cardiac computed tomography: Computed tomography was performed in a 64-slice scanner (Aquillion 64, Toshiba, Ottawara, Japan). Axial slices of 3 mm thickness with 3 mm table-feed were acquired at 70% of R-R interval with prospective ECG triggering. Coronary artery calcification was defined as a minimum of 3 contiguous pixels with a peak Hounsfield unit density > 130. Coronary artery calcifications were scored by a certified radiologist. The Agatston score was used to express the value of CAC.

ELIGIBILITY:
Inclusion Criteria:

* Aged of 80 years or over

Exclusion Criteria:

* Manifested atherosclerotic disease (MI, stroke or peripheral arterial disease) according to medical evaluation, electrocardiogram and echocardiogram
* Functional dependence or institutionalization
* Cognitive impairment assessed by mini-mental state examination (< 13 points)
* Use of any anti-inflammatory in the last 30 days
* Current or previous diagnosis of neoplastic or immune inflammatory disease
* Chronic obstructive pulmonary disease
* Glomerular filtration rate < 25 mL/min/1.73 m2
* Hepatic disease (ALT or AST ≥ 1.5 upper reference limit)
* Chronic infectious disease (≥ 3 months)
* Left ventricular ejection fraction < 50% on echocardiography
* Manifested neoplasia at admission or until the first year after enrollment

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Non-institutionalized outpatients under preventive care were voluntarily enrolled into the study. Participants were aged of 80 years or over, have never manifested myocardial infarction, stroke or peripheral arterial disease.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2008-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 1 year

SECONDARY OUTCOMES:
Major cardiovascular events | 2 years
  Sudden cardiac death (unrelated to trauma, unexpected, and occurring in less than six hours after onset of symptoms), fatal MI (any death preceded by MI) or non-fatal MI.

CONTACTS AND LOCATIONS:
Overall Officials: Andrei C Sposito, Ph.D., Principal Investigator — University of Campinas
Locations (2):
- Brazil (2):
  - Biocárdios - Instituto de Cardiologia, Brasília, Federal District
  - University of Campinas, Campinas, São Paulo

REFERENCES:
- [Background] Freitas WM, Quaglia LA, Santos SN, de Paula RC, Santos RD, Blaha M, Rivera JJ, Cury R, Blumenthal R, Nadruz-Junior W, Agatston A, Figueiredo VN, Nasir K, Sposito AC; Brazilian Study on Healthy Aging. Low HDL cholesterol but not high LDL cholesterol is independently associated with subclinical coronary atherosclerosis in healthy octogenarians. Aging Clin Exp Res. 2015 Feb;27(1):61-7. doi: 10.1007/s40520-014-0249-4. Epub 2014 Jun 7. PMID 24906678
- [Background] Henriques AD, Tonet-Furioso AC, Machado-Silva W, Freitas WM, Quaglia LA, Santos SN, Cordova C, Sposito AC, Nobrega OT; Brazilian Study on Healthy Aging Group. Apoliprotein E genotype is associated with apoliprotein B plasma levels but not with coronary calcium score in very elderly individuals in primary care setting. Gene. 2014 Apr 15;539(2):275-8. doi: 10.1016/j.gene.2014.01.077. Epub 2014 Feb 12. PMID 24530308
- [Background] Souza VC, Freitas WM, Quaglia LA, Santos SN, Cordova C, Sposito AC, Nobrega OT. Osteopontin in bone mineral density of very old Brazilians. J Bone Miner Metab. 2013 Jul;31(4):449-54. doi: 10.1007/s00774-013-0425-1. Epub 2013 Mar 21. PMID 23515922
- [Background] Costa AP, de Paula RC, Carvalho GF, Araujo JP, Andrade JM, de Almeida OL, de Faria EC, Freitas WM, Coelho OR, Ramires JA, Quinaglia e Silva JC, Sposito AC; Brasilia Heart Study Group. High sodium intake adversely affects oxidative-inflammatory response, cardiac remodelling and mortality after myocardial infarction. Atherosclerosis. 2012 May;222(1):284-91. doi: 10.1016/j.atherosclerosis.2012.02.037. Epub 2012 Mar 3. PMID 22436606
- [Background] Freitas WM, Quaglia LA, Santos SN, Soares AA, Japiassu AV, Boaventura V, dos Santos Barros E, Cordova C, Nobrega OT, Sposito AC. Association of systemic inflammatory activity with coronary and carotid atherosclerosis in the very elderly. Atherosclerosis. 2011 May;216(1):212-6. doi: 10.1016/j.atherosclerosis.2011.01.040. Epub 2011 Feb 2. PMID 21316055
- [Derived] de Azevedo Filho ER, Koeche C, Bueno FF, de Toledo O, Alves VP, da Silva HS, Moraes CF, Freitas WM, Campos-Staffico AM, de Carvalho LSF. Unraveling the intertwined threads of insomnia and sarcopenia in cognitive and functional impairment in octogenarians. BMC Geriatr. 2025 Nov 7;25(1):868. doi: 10.1186/s12877-025-06398-3. PMID 41204176